CLINICAL TRIAL: NCT03628716
Title: A Phase 2, Multicenter, Single-Arm Trial of CV301 in Combination With PD-1/L1 Blockade in Patients With Locally Advanced or Metastatic Urothelial Bladder Cancer
Brief Title: CV301 Combined With PD-1/L1 Blockade in Patients With Locally Advanced or Metastatic Urothelial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV301-BLD-001
Record Dates: First submitted 2018-08-03; First posted 2018-08-14 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CV301 + Atezolizumab (Experimental): Subject receiving combination treatment with CV301 + Atezolizumab
  Interventions: Biological: CV301; Biological: Atezolizumab

INTERVENTIONS:
Biological: CV301 — Prime with MVA-BN-CV301 (nominal titer 1.6 x 10^9 Inf.U) given subcutaneously (SC) on Day 1 and Day 22. One dose = four 0.5 mL injections. One injection = nominal titer 4 x 10^8 Inf.U in 0.5 mL.
  Boost with FPV-CV301 (nominal titer of 1 × 10^9 Inf.U in 0.5 mL, given SC every 21 days for 4 doses (on days 43, 64, 85, and 106), followed by boosts every 6 weeks until 6 months on trial (i.e., days 148 and 190), then every 12 weeks until completion of 2 years. One dose = one 0.5 mL injection.
Biological: Atezolizumab — Atezolizumab fixed dose of 1200 mg intravenous on Day 1 of each 21-day cycle

SUMMARY:
This is a Phase 2, single-arm, multi-institutional clinical trial designed to study the combination of CV301 with atezolizumab in the first-line treatment of UC not eligible for cisplatin-containing chemotherapy (Cohort 1) and in the second-line treatment of UC previously treated with standard first-line cisplatin-based chemotherapy (Cohort 2).

DETAILED DESCRIPTION:
This is a Phase 2, single-arm, multi-institutional clinical trial designed to study the combination of CV301 with atezolizumab in the first-line treatment of UC not eligible for cisplatin-containing chemotherapy (Cohort 1) and in the second-line treatment of UC previously treated with standard first-line cisplatin-based chemotherapy (Cohort 2). The trial will be performed using an optimal two-stage design within each cohort.

Stage 1, Cohort 1: Enroll 14 subjects. If objective response is not achieved in at least four patients, the cohort will be stopped for futility. If objective response is achieved in at least four subjects, the cohort will proceed to stage 2. If any patient is not evaluable for the primary endpoint, the patient may be replaced.

Stage 1, Cohort 2: Enroll 13 subjects. If objective response is not achieved in at least three patients, the cohort will be stopped for futility. If objective response is achieved in at least three subjects, the cohort will proceed to stage 2. If any patient is not evaluable for the primary endpoint, the patient may be replaced.

Stage 2, Cohort 1: Enroll an additional 19 subjects. If any patient is not evaluable for the primary endpoint, the patient may be replaced until a total of 33 patients are evaluable for the primary endpoint.

Stage 2, Cohort 2: Enroll an additional 22 subjects. If any patient is not evaluable for the primary endpoint, the patient may be replaced until a total of 35 patients are evaluable for the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at date of ICF signature having the ability to comply with protocol.
2. Histologically or cytologically documented locally advanced (T4b, any N; or any T, N 2-3) or metastatic (M1, Stage IV; or metastatic recurrence after locoregional treatment) UC (including renal pelvis, ureters, urinary bladder, urethra)

   1. Patients with mixed histologies were required to have a dominant transitional cell pattern.
   2. Locally advanced bladder cancer that was inoperable on the basis of involvement of the pelvic sidewall or adjacent viscera (clinical stage T4b) or bulky nodal metastasis (N2-N3).
3. Life expectancy ≥ 12 weeks.
4. Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions cannot be counted as target lesions unless there has been demonstrated progression in the lesion since radiotherapy and no other lesions are available for selection as target lesions.
5. Demonstrate adequate organ function.
6. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 5 months after the last dose of atezolizumab.
7. Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks preferred) or 10-15 unstained slides, with an associated pathology report.

   For Cohort 1:
8. Untreated with chemotherapy
9. Have at least one of the following:

   1. ECOG (Eastern Cooperative Oncology Group) performance status of 2.
   2. Glomerular filtration rate calculated as creatinine clearance (Cockroft-Gault formula) of ≥20 mL/min and less than 60 mL/min
   3. Hearing loss or neuropathy of any cause Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2

   For Cohort 2:
10. Disease progression during or following treatment with at least one platinum-containing regimen (e.g., GC, MVAC, CarboGem, carboplatin-paclitaxel) for inoperable locally advanced or metastatic urothelial carcinoma or disease recurrence, as defined by:

    1. Regimen is defined as patients receiving at least one cycle of a platinum-containing regimen with response assessment. Patients who received one cycle of a platinum-containing regimen but discontinued due to toxicity are also eligible.
    2. Patients who received prior adjuvant/neoadjuvant chemotherapy and progressed within 12 months of treatment with a platinum-containing adjuvant/neoadjuvant regimen are considered as second-line patients.
11. ECOG (Eastern Cooperative Oncology Group) performance status of < 2
12. Calculated creatinine clearance (Cockroft-Gault formula) of ≥20 mL/min

Exclusion Criteria:

1. Any approved anti-cancer therapy, including chemotherapy, within 3 weeks prior to initiation of trial treatment; the following exceptions are allowed:

   1. Palliative radiotherapy for bone metastases or non-target soft tissue lesions completed >7 days prior to baseline imaging.
   2. Hormone-replacement therapy or oral contraceptives.
2. Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to screening given that all AEs related to prior treatment have resolved to baseline or Grade 1.
3. Active central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments or Leptomeningeal disease.
4. Uncontrolled tumor-related pain:

   1. Patients requiring pain medication must be on a stable regimen at trial entry.
   2. Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to trial entry.
   3. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not currently associated with spinal cord compression) could be considered for loco-regional therapy if appropriate prior to enrollment.
5. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

   a. Patients with indwelling catheters (e.g., PleurX) are allowed.
6. Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium or Ca >12 mg/dL or corrected serum calcium >ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab:

   1. Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who did not have a history of clinically significant hypercalcemia are eligible.
   2. Patients who are receiving denosumab prior to enrollment have to be willing and eligible to receive a bisphosphonate instead while in the trial.
7. Malignancies other than urothelial carcinoma within 3 years prior to Day 1, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and no intent for further treatment or incidental prostate cancer (T1/T2b, Gleason score ≤7 undergoing active surveillance and treatment naive).
8. Pregnant and lactating women.
9. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, or aminoglycoside antibiotics or egg products, poxvirus-based vaccinations, or beef or bovine meat.
10. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation.
11. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, granulomatosis with polyangiitis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    1. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this trial.
    2. Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen are eligible for this trial.
    3. Patients with history of vitiligo and controlled psoriasis are eligible for the trial.
12. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan

    a. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
13. Positive test for Human Immunodeficiency Virus (HIV).
14. Patients with active hepatitis B virus (HBV; chronic or acute, defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C virus (HCV)

    1. Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HbsAg, negative polymerase chain reaction (PCR) for HBV) are eligible. HBV Deoxyribonucleic Acid (DNA) PCR must be obtained in these patients prior to Day 1.
    2. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV Ribonucleic Acid (RNA) prior to enrollment.
15. Active tuberculosis.
16. Signs or symptoms clinically significant of infection within 2 weeks prior to Day 1.
17. Received therapeutic oral or intravenous (IV) antibiotics within 1 week prior to Day 1

    a. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
18. Significant cardiovascular disease, which includes but is not limited to New York Heart Association (NYHA) Heart Failure Class II or greater, myocardial infarction within the previous 3 months, unstable arrhythmias, unstable angina.

    a. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% on a stable medical regimen that was optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate, are eligible.
19. Major surgical procedure other than for diagnosis within 28 days prior to Day 1 or anticipation of need for a major surgical procedure during the course of the trial.
20. Prior allogeneic stem cell or solid organ transplant.
21. Administration of a live, attenuated vaccine within 4 weeks before Day 1 or anticipation that such a live attenuated vaccine would be required during the trial

    a. Influenza vaccination may be given during influenza season only (approximately October to March). Patients cannot receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Day 1 or at any time during the trial.
22. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or that could affect the interpretation of the results or render the patient at high risk from treatment complications.
23. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
24. Treatment with systemic immunostimulatory agents (including but not limited to IFNs, interleukin [IL]-2) within 6 weeks or five half-lives of the drug, whichever was shorter, prior to Day 1.
25. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial

    a. Patients who receive acute, low-dose, systemic corticosteroid medications (e.g., a one-time dose of dexamethasone for nausea) or for prevention of hypersensitivity reactions to contrast agents may be enrolled in the trial.
26. The use of inhaled, nasal, ophthalmic, intra-articular, auricular or topical corticosteroids, physiologic replacement doses of glucocorticoids (i.e., for adrenal insufficiency), and mineralocorticoids (e.g. Fludrocortisone for adrenal insufficiency) is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CV301 + Atezolizumab (Cohort 1): Cohort 1 - Combination of CV301 with atezolizumab in the first-line treatment of urothelia cancer not eligible for cisplatin-containing chemotherapy
- CV301 + Atezolizumab (Cohort 2): Cohort 2 - Combination of CV301 with atezolizumab in the second-line treatment of urothelia cancer previously treated with standard first-line cisplatin-based chemotherapy
Period: Overall Study
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Started | 19 | 24
Completed | 0 | 1
Not Completed | 19 | 23
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 15 | 20
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Study Terminated by Sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Groups:
- Total: Total of all reporting groups
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2) | Total
Number analyzed (Participants) | 19 | 24 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 8 | 8
  >=65 years | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.0 (5.97) | 66.8 (10.99) | 72.2 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 16 | 19 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 23 | 41
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 24 | 43
ECOG Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status scales/grades are used to assess how a patient's disease is progressing. Grade 0=Fully active, able to carry on all pre-disease performance without restriction. Grade 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. Grade 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Grade 3=Capable of only limited self-care. Grade 4=Completely disabled. Grade 5=Dead.
  Participants
    Grade 0 | 10 | 12 | 22
    Grade 1 | 8 | 11 | 19
    Grade >=2 | 1 | 1 | 2
Primary Tumor Site [Count of Participants; unit: Participants]
  Renal Pelvis | 4 | 0 | 4
  Ureter | 1 | 0 | 1
  Urethra | 1 | 3 | 4
  Urinary Bladder | 13 | 21 | 34
Stage at Diagnosis [Count of Participants; unit: Participants] — Stage refers to the extent of cancer. Stage I=Early-stage or Localized (T1, N0, M0). Stage II=Localized (T2a or T2b, N0, M0). Stage III=Regional Spread (T3a, T3b, or T4a N0, M0). Stage IV=Distant Spread (T4b, N0, M0 or Any T, N1 to N3, M0 or Any T, Any N, M1).
  Participants
    Stage I | 7 | 3 | 10
    Stage II | 1 | 1 | 2
    Stage III | 4 | 4 | 8
    Stage IV | 7 | 16 | 23
T Category [Count of Participants; unit: Participants] — TX=Main tumor cannot be assessed due to lack of information. T0=No evidence of a primary tumor. Ta=Non-invasive papillary carcinoma. Tis=Non-invasive flat carcinoma. T1=Tumor has grown from the layer of cells lining the bladder into the connective tissue below. T2a=Tumor has grown into the outer half of the muscle layer. T3a=Spread to fatty tissue can only be seen by using microscope. T3b=Spread to fatty tissue that is large enough to be seen. T4a=Tumor has spread to the stroma of the prostate or to the uterus and/or vagina. T4b=Tumor has spread into the pelvic wall or abdominal wall.
  Participants
    TX | 4 | 4 | 8
    T0 | 0 | 0 | 0
    Ta | 3 | 2 | 5
    Tis | 1 | 1 | 2
    T1 | 4 | 7 | 11
    T2a | 0 | 1 | 1
    T2b | 2 | 1 | 3
    T3a | 2 | 1 | 3
    T3b | 2 | 4 | 6
    T4a | 0 | 2 | 2
    T4b | 1 | 1 | 2
N Category [Count of Participants; unit: Participants] — NX=Regional lymph nodes 8 cannot be assessed due to lack of information. N0=There is no regional lymph node spread. N1=Cancer has spread to a single lymph node in the true pelvis. N2=Cancer has spread to 2 or more lymph nodes in the true pelvis. N3=Cancer has spread to lymph nodes along the common iliac artery.
  Participants
    NX | 3 | 3 | 6
    N0 | 11 | 10 | 21
    N1 | 3 | 3 | 6
    N2 | 1 | 7 | 8
    N3 | 1 | 1 | 2
M Category [Count of Participants; unit: Participants] — M0=There are no signs of 9 distant spread. M1=Cancer has spread to distant parts of the body.
  Participants
    M0 | 10 | 10 | 20
    M1 | 8 | 14 | 22
    Not Reported | 1 | 0 | 1
Baseline PD-L1 Expression Tumor Proportion Score [Count of Participants; unit: Participants] — Programmed death ligand 1 (PD-L1) expression Tumor Proportion Score (TPS) is the percentage of viable tumor cells showing partial or complete membrane staining. No PD-L1 expression if TPS score is less than 1%.
  Participants
    <1% | 3 | 2 | 5
    >=1%-1<10% | 0 | 2 | 2
    >=10% | 0 | 0 | 0
    Not Applicable | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is the proportion of subjects in the analysis population with a Complete Response (CR) or Partial Response (PR) based on best overall RECIST v1.1 evaluations as performed by the investigator. According to RECIST v1.1, the sum of the longest diameters of non-nodal target lesions and short axis of nodal target lesions are used to evaluate tumor response. Maximum of 2 target lesions per organ and 5 target lesions are used for the measurement. CR means disappearance of all known disease, confirmed at 4 week, lymph nodes must be < 10 mm short axis. PR means >=30% decrease from baseline measurement, confirmed at 4 week.
Time Frame: up to 24 months
Population: Full Analysis Set subjects with objective response
Measure: Count of Participants; unit: Participants
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
Participants | 1 | 2

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The time interval from first treatment to objective tumor progression or death of any cause. Subjects without death or progression are censored at the date when the last assessment determined a lack of progression. The time interval from first vaccination to death of any cause, up to 4 years for each subject or discontinuation of the study by sponsor.
Time Frame: The time from day of first treatment to the start of disease progression or death, whichever occurs first, or the last assessment date if there is a lack of progression, up to 24 months for each subject or discontinuation of the study by sponsor.
Population: Full Analysis Set subjects with objective response
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
Months | 2 [1.68 to 2.10] | 1.95 [1.87 to 2.07]

3. Secondary Outcome: Overall Survival (OS)
Description: Time interval from first treatment to death of any cause. Subjects are censored at their date of last contact if they did not meet the survival endpoint by the outcome measure time frame.
Time Frame: The time interval from first vaccination to death of any cause, up to 24 months for each subject or discontinuation of the study by sponsor.
Population: Full Analysis Set: consists of all subjects taking any amount of trial vaccine
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
Months | 13.8 [2.37 to NA] — It is NA because it is not evaluable. There are insufficient subjects with events. | 8.13 [4.30 to NA] — It is NA because it is not evaluable. There are insufficient subjects with events.

4. Secondary Outcome: Duration of Response
Description: The time from objective response (CR or PR, whichever comes first) to investigator assessed progression using RECIST v1.1 or death
Time Frame: up to 24 months
Population: Full Analysis Set subjects with objective response
Measure: Median (90% Confidence Interval); unit: Months
Groups:
- CV301 + Atezolizumab (Cohort 1): Combination of CV301 with atezolizumab in the first-line treatment of urothelia cancer not eligible for cisplatin-containing chemotherapy
- CV301 + Atezolizumab (Cohort 2): Combination of CV301 with atezolizumab in the second-line treatment of urothelia cancer previously treated with standard first-line cisplatin-based chemotherapy
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 1 | 2
Months | NA [NA to NA] — It is NA because it is not evaluable. There are insufficient subject with events for estimation. | NA [NA to NA] — It is NA because it is not evaluable. There are insufficient subject with events for estimation.

5. Secondary Outcome: Treatment-Emergent Adverse Events
Description: An Overall Summary of Subjects with any Treatment-Emergent Adverse Events (TEAEs) and TEAEs Categories. TEAEs Categories include Related Adverse Events, >=Grade 3 Adverse Events, Related >= Grade 3 Adverse Events, Serious Adverse Events, Related Serious Adverse Events, Adverse Events of Special Interest and Related Adverse Events of Special Interest. TEAEs are considered as related when the investigator-assessed relationship of the corresponding trial treatment is "possible", "probable", "definite" or missing. Per CTCAE v5, Grade 1=Mild; asymptomatic or mild symptoms. Grade 2=Moderate; minimal, local or noninvasive intervention indicated. Grade 3=Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. Grade 4=Life-threatening consequences; urgent intervention indicated. Grade 5=Death related to AE. Immune Mediated Adverse Events (IMAE) and Cardiac events are considered AESIs.
Time Frame: up to 24 months
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
Participants
  Treatment Emergent Adverse Events | 19 | 24
  Related Adverse Events | 16 | 21
  >= Grade 3 Adverse Events | 10 | 12
  Related >= Grade 3 Adverse Events | 5 | 4
  Serious Adverse Events | 7 | 5
  Related Serious Adverse Events | 0 | 1
  Adverse Events of Special Interest | 1 | 1
  Related Adverse Events of Special Interest | 0 | 1

6. Secondary Outcome: Toxicity Grade Shift From Baseline in Laboratory Results
Description: Toxicity grades are based on CTCAE v5 scales for hematology and chemistry laboratory parameters. Grade 0=Normal, Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 5=Life-threatening, and Grade 5=Death. Toxicity grade shift is defined to evaluate categorical changes from baseline results to post-treatment results with respect to dichotomized CTCAE v5 grading value (<= Grade 2, >= Grade 3).
Time Frame: Overall Study up to 24 months
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
Participants
  Eosinophils <= Grade 2: number analyzed (Participants) | 18 | 24
  Eosinophils <= Grade 2 | 18 | 24
  Eosinophils >= Grade 3: number analyzed (Participants) | 18 | 24
  Eosinophils >= Grade 3 | 0 | 0
  Hemoglobin <= Grade 2: number analyzed (Participants) | 18 | 24
  Hemoglobin <= Grade 2 | 18 | 24
  Hemoglobin >= Grade 3: number analyzed (Participants) | 18 | 24
  Hemoglobin >= Grade 3 | 0 | 0
  Leukocytes <= Grade 2: number analyzed (Participants) | 18 | 24
  Leukocytes <= Grade 2 | 18 | 24
  Leukocytes >= Grade 3: number analyzed (Participants) | 18 | 24
  Leukocytes >= Grade 3 | 0 | 0
  Lymphocytes <= Grade 2: number analyzed (Participants) | 18 | 24
  Lymphocytes <= Grade 2 | 16 | 22
  Lymphocytes >= Grade 3: number analyzed (Participants) | 18 | 24
  Lymphocytes >= Grade 3 | 2 | 2
  Neutrophils <= Grade 2: number analyzed (Participants) | 18 | 24
  Neutrophils <= Grade 2 | 18 | 24
  Neutrophils >= Grade 3: number analyzed (Participants) | 18 | 24
  Neutrophils >= Grade 3 | 0 | 0
  Platelets <= Grade 2: number analyzed (Participants) | 18 | 24
  Platelets <= Grade 2 | 18 | 24
  Platelets >= Grade 3: number analyzed (Participants) | 18 | 24
  Platelets >= Grade 3 | 0 | 0
  Alanine Aminotransferase <= Grade 2: number analyzed (Participants) | 18 | 24
  Alanine Aminotransferase <= Grade 2 | 18 | 24
  Alanine Aminotransferase >= Grade 3: number analyzed (Participants) | 18 | 24
  Alanine Aminotransferase >= Grade 3 | 0 | 0
  Albumin <= Grade 2: number analyzed (Participants) | 18 | 24
  Albumin <= Grade 2 | 18 | 24
  Albumin >= Grade 3: number analyzed (Participants) | 18 | 24
  Albumin >= Grade 3 | 0 | 0
  Alkaline Phosphatase <= Grade 2: number analyzed (Participants) | 18 | 24
  Alkaline Phosphatase <= Grade 2 | 18 | 24
  Alkaline Phosphatase >= Grade 3: number analyzed (Participants) | 18 | 24
  Alkaline Phosphatase >= Grade 3 | 0 | 0
  Amylase <= Grade 2: number analyzed (Participants) | 18 | 24
  Amylase <= Grade 2 | 17 | 24
  Amylase >= Grade 3: number analyzed (Participants) | 18 | 24
  Amylase >= Grade 3 | 1 | 0
  Aspartate Aminotransferase <= Grade 2: number analyzed (Participants) | 18 | 24
  Aspartate Aminotransferase <= Grade 2 | 18 | 24
  Aspartate Aminotransferase >= Grade 3: number analyzed (Participants) | 18 | 24
  Aspartate Aminotransferase >= Grade 3 | 0 | 0
  Bicarbonate <= Grade 2: number analyzed (Participants) | 18 | 24
  Bicarbonate <= Grade 2 | 18 | 24
  Bicarbonate >= Grade 3: number analyzed (Participants) | 18 | 24
  Bicarbonate >= Grade 3 | 0 | 0
  Bilirubin <= Grade 2: number analyzed (Participants) | 18 | 24
  Bilirubin <= Grade 2 | 17 | 24
  Bilirubin >= Grade 3: number analyzed (Participants) | 18 | 24
  Bilirubin >= Grade 3 | 1 | 0
  Calcium <= Grade 2: number analyzed (Participants) | 18 | 24
  Calcium <= Grade 2 | 18 | 24
  Calcium >= Grade 3: number analyzed (Participants) | 18 | 24
  Calcium >= Grade 3 | 0 | 0
  Creatinine <= Grade 2: number analyzed (Participants) | 18 | 24
  Creatinine <= Grade 2 | 16 | 24
  Creatinine >= Grade 3: number analyzed (Participants) | 18 | 24
  Creatinine >= Grade 3 | 2 | 0
  Glucose <= Grade 2: number analyzed (Participants) | 18 | 24
  Glucose <= Grade 2 | 18 | 24
  Glucose >= Grade 3: number analyzed (Participants) | 18 | 24
  Glucose >= Grade 3 | 0 | 0
  Lactate Dehydrogenase <= Grade 2: number analyzed (Participants) | 18 | 24
  Lactate Dehydrogenase <= Grade 2 | 18 | 24
  Lactate Dehydrogenase >= Grade 3: number analyzed (Participants) | 18 | 24
  Lactate Dehydrogenase >= Grade 3 | 0 | 0
  Lipase <= Grade 2: number analyzed (Participants) | 18 | 24
  Lipase <= Grade 2 | 15 | 23
  Lipase >= Grade 3: number analyzed (Participants) | 18 | 24
  Lipase >= Grade 3 | 3 | 1
  Potassium <= Grade 2: number analyzed (Participants) | 18 | 24
  Potassium <= Grade 2 | 18 | 24
  Potassium >= Grade 3: number analyzed (Participants) | 18 | 24
  Potassium >= Grade 3 | 0 | 0
  Sodium <= Grade 2: number analyzed (Participants) | 18 | 24
  Sodium <= Grade 2 | 18 | 22
  Sodium >= Grade 3: number analyzed (Participants) | 18 | 24
  Sodium >= Grade 3 | 0 | 2
  Thyrotropin <= Grade 2: number analyzed (Participants) | 13 | 18
  Thyrotropin <= Grade 2 | 13 | 18
  Thyrotropin >= Grade 3: number analyzed (Participants) | 13 | 18
  Thyrotropin >= Grade 3 | 0 | 0
  Urate <= Grade 2: number analyzed (Participants) | 18 | 24
  Urate <= Grade 2 | 12 | 21
  Urate >= Grade 3: number analyzed (Participants) | 18 | 24
  Urate >= Grade 3 | 6 | 3

7. Secondary Outcome: Vital Signs Results - Pulse Rate
Description: Vital signs results assessed throughout the study.
Time Frame: Overall study up to 24 months
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
beats per minute
  Baseline | 76.4 (13.41) | 75.3 (15.31)
  Week 4: number analyzed (Participants) | 18 | 24
  Week 4 | 72.7 (11.49) | 79.4 (17.61)
  Week 7: number analyzed (Participants) | 13 | 19
  Week 7 | 70.2 (12.06) | 76.5 (15.56)
  Week 10: number analyzed (Participants) | 10 | 18
  Week 10 | 66.8 (8.84) | 79.5 (17.06)
  Week 13: number analyzed (Participants) | 8 | 7
  Week 13 | 73.6 (11.45) | 75.0 (18.46)
  Week 16: number analyzed (Participants) | 8 | 7
  Week 16 | 66.5 (5.58) | 76.7 (15.74)
  Week 19: number analyzed (Participants) | 5 | 6
  Week 19 | 66.4 (11.01) | 76.2 (17.49)
  Week 22: number analyzed (Participants) | 5 | 6
  Week 22 | 72.2 (16.95) | 71.7 (18.04)
  Week 25: number analyzed (Participants) | 3 | 5
  Week 25 | 68.7 (17.56) | 83.0 (13.73)
  Week 28: number analyzed (Participants) | 3 | 5
  Week 28 | 57.3 (5.51) | 83.4 (23.95)
  Week 31: number analyzed (Participants) | 3 | 3
  Week 31 | 64.0 (11.14) | 86.0 (14.73)
  Week 34: number analyzed (Participants) | 3 | 3
  Week 34 | 67.3 (13.58) | 74.7 (8.08)
  Week 37: number analyzed (Participants) | 2 | 3
  Week 37 | 76.5 (30.41) | 80.0 (10.15)
  Week 40: number analyzed (Participants) | 3 | 3
  Week 40 | 67.0 (14.11) | 84.7 (13.32)
  Week 43: number analyzed (Participants) | 1 | 3
  Week 43 | 68.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 subjects were analyzed. | 85.3 (17.21)
  Week 46: number analyzed (Participants) | 1 | 3
  Week 46 | 69.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 91.7 (11.37)
  Week 49: number analyzed (Participants) | 1 | 3
  Week 49 | 93.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 80.0 (6.93)
  Week 52: number analyzed (Participants) | 1 | 3
  Week 52 | 75.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 94.7 (17.5)
  Week 55: number analyzed (Participants) | 1 | 2
  Week 55 | 79.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 74.0 (7.07)
  Week 58: number analyzed (Participants) | 0 | 2
  Week 58 |  | 75.5 (0.71)
  Week 61: number analyzed (Participants) | 1 | 2
  Week 61 | 68.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 77.5 (10.61)
  Week 64: number analyzed (Participants) | 1 | 2
  Week 64 | 81.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 81.0 (1.41)
  Week 67: number analyzed (Participants) | 0 | 2
  Week 67 |  | 81.0 (2.83)
  Week 70: number analyzed (Participants) | 1 | 2
  Week 70 | 80.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 73.0 (5.66)
  Week 73: number analyzed (Participants) | 0 | 2
  Week 73 |  | 72.0 (9.90)
  Week 76: number analyzed (Participants) | 0 | 2
  Week 76 |  | 85.0 (5.66)
  Week 79: number analyzed (Participants) | 1 | 2
  Week 79 | 77.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 76.0 (12.73)
  Week 82: number analyzed (Participants) | 0 | 1
  Week 82 |  | 73.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 85: number analyzed (Participants) | 1 | 1
  Week 85 | 80.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 66.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 88: number analyzed (Participants) | 0 | 1
  Week 88 |  | 77.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 91: number analyzed (Participants) | 1 | 1
  Week 91 | 58.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 69.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 94: number analyzed (Participants) | 1 | 1
  Week 94 | 83.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 84.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 97: number analyzed (Participants) | 1 | 1
  Week 97 | 63.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 81.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 100: number analyzed (Participants) | 1 | 1
  Week 100 | 64.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 93.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.

8. Secondary Outcome: Vital Signs Results - System Blood Pressure
Description: Vital signs results assessed throughout the study.
Time Frame: Overall study up to 24 months
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
mmHg
  Baseline | 127.0 (18.72) | 129.9 (16.15)
  Week 4: number analyzed (Participants) | 18 | 24
  Week 4 | 121.3 (16.43) | 123.2 (13.29)
  Week 7: number analyzed (Participants) | 13 | 19
  Week 7 | 135.1 (20.35) | 125.9 (11.29)
  Week 10: number analyzed (Participants) | 10 | 18
  Week 10 | 130.0 (18.13) | 126.5 (11.75)
  Week 13: number analyzed (Participants) | 8 | 7
  Week 13 | 129.9 (12.19) | 129.7 (7.5)
  Week 16: number analyzed (Participants) | 8 | 7
  Week 16 | 133.5 (17.88) | 127.4 (10.16)
  Week 19: number analyzed (Participants) | 5 | 6
  Week 19 | 141.2 (17.91) | 113.7 (12.08)
  Week 22: number analyzed (Participants) | 5 | 6
  Week 22 | 139.2 (36.08) | 121.0 (11.49)
  Week 25: number analyzed (Participants) | 3 | 5
  Week 25 | 146.0 (27.06) | 129.4 (12.54)
  Week 28: number analyzed (Participants) | 3 | 5
  Week 28 | 139.3 (35.8) | 123.8 (11.69)
  Week 31: number analyzed (Participants) | 3 | 3
  Week 31 | 134.7 (6.66) | 118.7 (3.79)
  Week 34: number analyzed (Participants) | 3 | 3
  Week 34 | 130.3 (8.74) | 124.3 (4.51)
  Week 37: number analyzed (Participants) | 2 | 3
  Week 37 | 140.0 (1.41) | 138.0 (19.92)
  Week 40: number analyzed (Participants) | 3 | 3
  Week 40 | 140.0 (20.42) | 111.0 (15.87)
  Week 43: number analyzed (Participants) | 1 | 3
  Week 43 | 141.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 129.3 (11.72)
  Week 46: number analyzed (Participants) | 1 | 3
  Week 46 | 177.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 132.7 (3.79)
  Week 49: number analyzed (Participants) | 1 | 3
  Week 49 | 150.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 127.7 (15.04)
  Week 52: number analyzed (Participants) | 1 | 3
  Week 52 | 154.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 120.3 (17.79)
  Week 55: number analyzed (Participants) | 1 | 2
  Week 55 | 149.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 139.0 (4.24)
  Week 58: number analyzed (Participants) | 0 | 2
  Week 58 |  | 134.0 (2.83)
  Week 61: number analyzed (Participants) | 1 | 2
  Week 61 | 150.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 132.0 (9.9)
  Week 64: number analyzed (Participants) | 1 | 2
  Week 64 | 155.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 129.0 (1.41)
  Week 67: number analyzed (Participants) | 0 | 2
  Week 67 |  | 143.0 (8.49)
  Week 70: number analyzed (Participants) | 1 | 2
  Week 70 | 148.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 138.5 (10.61)
  Week 73: number analyzed (Participants) | 0 | 2
  Week 73 |  | 140.0 (11.31)
  Week 76: number analyzed (Participants) | 0 | 2
  Week 76 |  | 119.0 (26.87)
  Week 79: number analyzed (Participants) | 1 | 2
  Week 79 | 142.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 125.0 (1.41)
  Week 82: number analyzed (Participants) | 0 | 1
  Week 82 |  | 118.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 85: number analyzed (Participants) | 1 | 1
  Week 85 | 169.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 134.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 88: number analyzed (Participants) | 0 | 1
  Week 88 |  | 116.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 91: number analyzed (Participants) | 1 | 1
  Week 91 | 142.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 135.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 94: number analyzed (Participants) | 1 | 1
  Week 94 | 148.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 136.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 97: number analyzed (Participants) | 1 | 1
  Week 97 | 159.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 125.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 100: number analyzed (Participants) | 1 | 1
  Week 100 | 165.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 120.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.

9. Secondary Outcome: Vital Signs Results - Diastolic Blood Pressure
Description: Vital signs results assessed throughout the study.
Time Frame: Overall study up to 24 months
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
mmHg
  Baseline | 68.3 (8.39) | 74.4 (9.33)
  Week 4: number analyzed (Participants) | 18 | 24
  Week 4 | 67.4 (7.18) | 70.5 (9.08)
  Week 7: number analyzed (Participants) | 13 | 19
  Week 7 | 70.0 (8.42) | 71.8 (9.58)
  Week 10: number analyzed (Participants) | 10 | 18
  Week 10 | 71.3 (10.06) | 71.6 (8.75)
  Week 13: number analyzed (Participants) | 8 | 7
  Week 13 | 74.0 (8.43) | 73.0 (6.86)
  Week 16: number analyzed (Participants) | 8 | 7
  Week 16 | 70.4 (8.26) | 74.7 (8.67)
  Week 19: number analyzed (Participants) | 5 | 6
  Week 19 | 68.0 (5.34) | 68.8 (10.57)
  Week 22: number analyzed (Participants) | 5 | 6
  Week 22 | 72.6 (9.58) | 64.2 (10.82)
  Week 25: number analyzed (Participants) | 3 | 5
  Week 25 | 73.0 (6.08) | 73.8 (9.81)
  Week 28: number analyzed (Participants) | 3 | 5
  Week 28 | 64.3 (10.02) | 74.8 (5.89)
  Week 31: number analyzed (Participants) | 3 | 3
  Week 31 | 71.7 (7.51) | 76.0 (8.19)
  Week 34: number analyzed (Participants) | 3 | 3
  Week 34 | 67.3 (5.03) | 74.7 (2.52)
  Week 37: number analyzed (Participants) | 2 | 3
  Week 37 | 83.0 (1.41) | 81.0 (10.44)
  Week 40: number analyzed (Participants) | 3 | 3
  Week 40 | 68.0 (7.21) | 70.0 (8.72)
  Week 43: number analyzed (Participants) | 1 | 3
  Week 43 | 69.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 76.0 (1.00)
  Week 46: number analyzed (Participants) | 1 | 3
  Week 46 | 80.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 82.7 (3.21)
  Week 49: number analyzed (Participants) | 1 | 3
  Week 49 | 69.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 76.7 (3.51)
  Week 52: number analyzed (Participants) | 1 | 3
  Week 52 | 73.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 74.0 (10.00)
  Week 55: number analyzed (Participants) | 1 | 2
  Week 55 | 64.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 82.5 (9.19)
  Week 58: number analyzed (Participants) | 0 | 2
  Week 58 |  | 78.5 (4.95)
  Week 61: number analyzed (Participants) | 1 | 2
  Week 61 | 56.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 76.5 (7.78)
  Week 64: number analyzed (Participants) | 1 | 2
  Week 64 | 70.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 73.5 (3.54)
  Week 67: number analyzed (Participants) | 0 | 2
  Week 67 |  | 73.5 (0.71)
  Week 70: number analyzed (Participants) | 1 | 2
  Week 70 | 81.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 71.5 (2.12)
  Week 73: number analyzed (Participants) | 0 | 2
  Week 73 |  | 79.5 (14.85)
  Week 76: number analyzed (Participants) | 0 | 2
  Week 76 |  | 67.5 (4.95)
  Week 79: number analyzed (Participants) | 1 | 2
  Week 79 | 69.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 72.5 (2.12)
  Week 82: number analyzed (Participants) | 0 | 1
  Week 82 |  | 60.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 85: number analyzed (Participants) | 1 | 1
  Week 85 | 71.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 77.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 88: number analyzed (Participants) | 0 | 1
  Week 88 |  | 78.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 91: number analyzed (Participants) | 1 | 1
  Week 91 | 61.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 83.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 94: number analyzed (Participants) | 1 | 1
  Week 94 | 66.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 62.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 97: number analyzed (Participants) | 1 | 1
  Week 97 | 72.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 66.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 100: number analyzed (Participants) | 1 | 1
  Week 100 | 69.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 72.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.

10. Secondary Outcome: Vital Signs Results - Temperature
Description: Vital signs results assessed throughout the study.
Time Frame: Overall study up to 24 months
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
Celsius
  Baseline | 36.58 (0.310) | 36.64 (0.239)
  Week 4: number analyzed (Participants) | 18 | 24
  Week 4 | 36.63 (0.218) | 36.57 (0.232)
  Week 7: number analyzed (Participants) | 13 | 19
  Week 7 | 36.60 (0.196) | 36.66 (0.292)
  Week 10: number analyzed (Participants) | 10 | 18
  Week 10 | 36.61 (0.166) | 36.51 (0.241)
  Week 13: number analyzed (Participants) | 8 | 7
  Week 13 | 36.57 (0.167) | 36.53 (0.327)
  Week 16: number analyzed (Participants) | 8 | 7
  Week 16 | 36.63 (0.191) | 36.62 (0.213)
  Week 19: number analyzed (Participants) | 5 | 6
  Week 19 | 36.68 (0.217) | 36.45 (0.367)
  Week 22: number analyzed (Participants) | 5 | 6
  Week 22 | 36.70 (0.316) | 36.44 (0.382)
  Week 25: number analyzed (Participants) | 3 | 4
  Week 25 | 36.61 (0.322) | 36.62 (0.320)
  Week 28: number analyzed (Participants) | 3 | 5
  Week 28 | 36.67 (0.153) | 36.72 (0.416)
  Week 31: number analyzed (Participants) | 3 | 3
  Week 31 | 36.75 (0.330) | 36.56 (0.161)
  Week 34: number analyzed (Participants) | 3 | 3
  Week 34 | 36.71 (0.013) | 36.65 (0.274)
  Week 37: number analyzed (Participants) | 2 | 3
  Week 37 | 36.84 (0.644) | 36.70 (0.213)
  Week 40: number analyzed (Participants) | 3 | 3
  Week 40 | 36.61 (0.379) | 37.17 (0.409)
  Week 43: number analyzed (Participants) | 1 | 3
  Week 43 | 36.80 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.86 (0.076)
  Week 46: number analyzed (Participants) | 1 | 3
  Week 46 | 36.80 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.59 (0.103)
  Week 49: number analyzed (Participants) | 1 | 3
  Week 49 | 36.70 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.79 (0.135)
  Week 52: number analyzed (Participants) | 1 | 3
  Week 52 | 36.90 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.72 (0.434)
  Week 55: number analyzed (Participants) | 1 | 2
  Week 55 | 36.40 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.53 (0.189)
  Week 58: number analyzed (Participants) | 0 | 2
  Week 58 |  | 36.66 (0.063)
  Week 61: number analyzed (Participants) | 1 | 2
  Week 61 | 36.60 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.53 (0.189)
  Week 64: number analyzed (Participants) | 1 | 2
  Week 64 | 36.70 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.64 (0.196)
  Week 67: number analyzed (Participants) | 0 | 2
  Week 67 |  | 36.60 (0.141)
  Week 70: number analyzed (Participants) | 1 | 2
  Week 70 | 36.80 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.51 (0.149)
  Week 73: number analyzed (Participants) | 0 | 2
  Week 73 |  | 36.35 (0.212)
  Week 76: number analyzed (Participants) | 0 | 2
  Week 76 |  | 36.76 (0.204)
  Week 79: number analyzed (Participants) | 1 | 2
  Week 79 | 37.10 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.12 (0.456)
  Week 82: number analyzed (Participants) | 0 | 1
  Week 82 |  | 36.70 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 85: number analyzed (Participants) | 1 | 1
  Week 85 | 36.20 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.30 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 88: number analyzed (Participants) | 0 | 1
  Week 88 |  | 36.60 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 91: number analyzed (Participants) | 1 | 1
  Week 91 | 36.40 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.30 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 94: number analyzed (Participants) | 1 | 1
  Week 94 | 36.60 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.10 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 97: number analyzed (Participants) | 1 | 1
  Week 97 | 36.70 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.60 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 100: number analyzed (Participants) | 1 | 1
  Week 100 | 36.90 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 36.60 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.

11. Secondary Outcome: Vital Signs Results - Respiratory Rate
Description: Vital signs results assessed throughout the study.
Time Frame: Overall study up to 24 months
Population: The Full Analysis Set consists of all subjects taking any amount of trial vaccine
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
Number analyzed (Participants) | 19 | 24
breaths per minute
  Baseline | 16.7 (0.99) | 16.7 (0.96)
  Week 4: number analyzed (Participants) | 18 | 24
  Week 4 | 17.0 (1.24) | 16.9 (1.23)
  Week 7: number analyzed (Participants) | 13 | 19
  Week 7 | 16.9 (1.04) | 16.6 (0.90)
  Week 10: number analyzed (Participants) | 10 | 18
  Week 10 | 16.6 (0.97) | 17.2 (1.69)
  Week 13: number analyzed (Participants) | 8 | 7
  Week 13 | 16.5 (0.93) | 16.0 (0.00)
  Week 16: number analyzed (Participants) | 8 | 7
  Week 16 | 17.0 (1.51) | 17.0 (2.24)
  Week 19: number analyzed (Participants) | 5 | 6
  Week 19 | 16.8 (1.10) | 15.3 (1.63)
  Week 22: number analyzed (Participants) | 5 | 6
  Week 22 | 16.8 (1.10) | 16.3 (0.82)
  Week 25: number analyzed (Participants) | 3 | 5
  Week 25 | 16.7 (1.15) | 16.0 (0.00)
  Week 28: number analyzed (Participants) | 3 | 5
  Week 28 | 17.3 (2.31) | 16.2 (0.45)
  Week 31: number analyzed (Participants) | 3 | 3
  Week 31 | 16.7 (1.15) | 16.0 (0.00)
  Week 34: number analyzed (Participants) | 3 | 3
  Week 34 | 18.0 (0.00) | 16.7 (1.15)
  Week 37: number analyzed (Participants) | 2 | 3
  Week 37 | 17.0 (1.41) | 15.3 (1.15)
  Week 40: number analyzed (Participants) | 3 | 3
  Week 40 | 16.7 (1.15) | 16.0 (0.00)
  Week 43: number analyzed (Participants) | 1 | 3
  Week 43 | 18.0 (NA) — It is NA because it is not evaluable. | 17.0 (1.73)
  Week 46: number analyzed (Participants) | 1 | 3
  Week 46 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 15.7 (0.58)
  Week 49: number analyzed (Participants) | 1 | 3
  Week 49 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 15.7 (0.58)
  Week 52: number analyzed (Participants) | 1 | 3
  Week 52 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 16.7 (1.15)
  Week 55: number analyzed (Participants) | 1 | 2
  Week 55 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 16.0 (0.00)
  Week 58: number analyzed (Participants) | 0 | 2
  Week 58 |  | 17.0 (1.41)
  Week 61: number analyzed (Participants) | 1 | 2
  Week 61 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 16.0 (0.00)
  Week 64: number analyzed (Participants) | 1 | 2
  Week 64 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 16.0 (0.00)
  Week 67: number analyzed (Participants) | 0 | 2
  Week 67 |  | 16.5 (0.71)
  Week 70: number analyzed (Participants) | 1 | 2
  Week 70 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 17.0 (1.41)
  Week 73: number analyzed (Participants) | 0 | 2
  Week 73 |  | 17.0 (1.41)
  Week 76: number analyzed (Participants) | 0 | 2
  Week 76 |  | 16.0 (0.00)
  Week 79: number analyzed (Participants) | 1 | 2
  Week 79 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 17.0 (1.41)
  Week 82: number analyzed (Participants) | 0 | 1
  Week 82 |  | 16.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 85: number analyzed (Participants) | 1 | 1
  Week 85 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 88: number analyzed (Participants) | 0 | 1
  Week 88 |  | 16.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 91: number analyzed (Participants) | 1 | 1
  Week 91 | 17.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 16.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 94: number analyzed (Participants) | 1 | 1
  Week 94 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 16.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 97: number analyzed (Participants) | 1 | 1
  Week 97 | 16.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.
  Week 100: number analyzed (Participants) | 1 | 1
  Week 100 | 18.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed. | 16.0 (NA) — It is NA because it is not evaluable. Standard deviation not calculated when <2 participants were analyzed.

ADVERSE EVENTS:
Time Frame: All Adverse events collected from the signing of inform consent form to 30 days after the last dose of trial product, if unrelated to trial product or non-serious, and all trial product-related SAEs and AESI collected through 100 days after the last dose of trial product, up to 24 months.
Description: All Adverse events collected from the signing of inform consent form to 30 days after the last dose of trial product, if unrelated to trial product or non-serious, and all trial product-related SAEs and AESI collected through 100 days after the last dose of trial product.
Arm/Group | CV301 + Atezolizumab (Cohort 1) | CV301 + Atezolizumab (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 11/19 | 15/24
Serious Adverse Events (participants affected / at risk) | 7/19 | 5/24
Other Adverse Events (participants affected / at risk) | 18/19 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CV301 + Atezolizumab (Cohort 1) (N=19) | CV301 + Atezolizumab (Cohort 2) (N=24)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CV301 + Atezolizumab (Cohort 1) (N=19) | CV301 + Atezolizumab (Cohort 2) (N=24)
Fatigue (General disorders) | 8 (9) | 8 (10)
Injection site pain (General disorders) | 2 (2) | 8 (14)
Pyrexia (General disorders) | 2 (2) | 6 (7)
Chills (General disorders) | 3 (4) | 4 (4)
Injection site erythema (General disorders) | 1 (1) | 6 (12)
Injection site swelling (General disorders) | 2 (2) | 4 (5)
Influenza like illness (General disorders) | 0 (0) | 4 (4)
Injection site mass (General disorders) | 0 (0) | 3 (7)
Injection site reaction (General disorders) | 1 (1) | 2 (2)
Injection site discomfort (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Infusion site uriticaria (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Injection site irritation (General disorders) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (7)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Adominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weaness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (5)
Kidney infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 3 (3) | 0 (0)
Lipase increased (Investigations) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Carbon dioxide decreased (Investigations) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Agreement entitles Bavarian Nordic to request the Institution(s) to delay their publication for a period of up to three (3) months from the date of the first submission to Bavarian Nordic.

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT03628716/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03628716/SAP_001.pdf